CLINICAL TRIAL: NCT00838461
Title: Multiple Ascending Dose Study of the Safety, Pharmacokinetics, and Pharmacodynamics of HSD-016 Administered Orally to Healthy Subjects
Brief Title: Study Evaluating the Safety, Pharmacokinetics (PK), and Pharmacodynamices (PD) of HSD-016
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 3248A1-1002
Record Dates: First submitted 2009-02-05; First posted 2009-02-06 (Estimated); Last update posted 2009-08-03 (Estimated); Status verified 2009-07

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — (R)-1,1,1-trifluoro-2-(3-((R)-4-(4-fluoro-2-(trifluoromethyl)phenyl)-2-methylpiperazin-1-ylsulfonyl)phenyl)propan-2-ol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): HSD-016
  Interventions: Drug: HSD-016
- 2 (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: HSD-016
  Arms: 1
Drug: placebo
  Arms: 2

SUMMARY:
This is intended to provide an initial safety assessment of HSD-016 and also to evaluate how the drug is absorbed and eliminated and its effect on the body in healthy subjects.

ELIGIBILITY:
Inclusion criteria:

1. Men or women of nonchildbearing potential aged 18 to 50 years.
2. Healthy as determined by investigator on the basis of medical history and physical examination, laboratory test results, and 12-lead ECG. 3. Nonsmoker or smoker of fewer than 10 cigarettes per day.

Exclusion criteria:

1. No history of thyroid abnormalities.
2. No presence or history of any disorder that may prevent the successful completion of the study.
3. No history of drug abuse.
4. No use of any systemic steroids for 3 months.
5. No history of claustrophobia.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2009-03; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Safety will be evaluated from reported AEs, scheduled physical, vital sign measurements, 12 lead ECGs, and clinical laboratory test results. | 3 months

SECONDARY OUTCOMES:
Levels of drug concentrations will be evaluated after receiving multiple doses of HSD-016 | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Chula Vista, California, United States